CLINICAL TRIAL: NCT03068572
Title: A Study on the Diagnosis of Minimal Change Esophagitis in Nonerosive Reflux Esophagitis and Gastroesophageal Reflux Disease Using Linked Color Imaging
Brief Title: Diagnostic Value of Linked Color Imaging for Minimal Change Esophagitis in Nonerosive Reflux Esophagitis and GERD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 307LCI-MCE
Record Dates: First submitted 2017-02-22; First posted 2017-03-03 (Actual); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Gastroesophageal Reflux Disease; Minimal Change Disease; Non-Reflux Esophagitis
Keywords: minimal change esophageal reflux disease diagnosis; Linked Color imaging; non-erosive reflux disease
MeSH Terms: conditions — Gastroesophageal Reflux; Nephrosis, Lipoid; Non-Erosive Reflux Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NERD group: 45 GERD patients without obviously abnormality were examined by conventional white-light endoscopy and then followed by Linked Color imaging(LCI) to evaluate minimal change esophagitis and observation agreement of Los Angeles classification system GERD patients with the absence of mucosal breaks at conventional endoscopy,and those patients was given standard or double dose of oral proton pump inhibitor (PPI) for 2 weeks to determine the efficacy of anti-secretory therapy (the so-called PPI test).The response to PPI treatment comprised the NERD group.
- Control group: 45 control patients were examined by white-light endoscopy and then followed by Linked Color imaging(LCI) to evaluate minimal change esophagitis and observation agreement of Los Angeles classification system,those subjects who had undergone endoscopy solely for the purpose of a health check-up at the same time of the study period

SUMMARY:
Linked color imaging(LCI),a new system for endoscopy modality,creates clear and bright endoscopic images by using short-wavelength narrow-band laser light combined with white laser light on the basis of magnifying blue laser imaging(BLI) technology.LCI makes red areas appear redder and white areas appear whiter.Thus,it is easier to recognize a slight difference in color of the mucosa.This is a study to assess the effectiveness of LCI for diagnosing esophageal minimal endoscopic lesions and Los Angeles classification system when compared to conventional white-light endoscopy (WLI).Gastroesophageal reflux disease(GERD) is a common disease that be defined as a condition which develops when the reflux of stomach contents cause troublesome symptoms and/or complications.Esophageal injury was classified according to the Los Angeles classification system,Non-erosive reflux disease(NERD) is defined by the presence of troublesome reflux-associated symptoms and the absence of mucosal breaks at endoscopy,which includes minimal change oesophagitis and no endoscopic abnormalities.LCI improved the visualization of the squamocolumnar junction (SCJ) by enhancing the contrast,mucosa minimal changes could be seen more easily and clearly with LCI than with standard white-light endoscopy.By comparing White-light endoscopy and LCI,it will show if there is any comparable advantage to using one or the other for lesion detection.

DETAILED DESCRIPTION:
This is a prospective study comparing the use of linked color imaging(LCI) versus standard white light for the detection of minimal change esophageal.Gastroesophageal reflux disease(GERD) is a common disease that be defined as a condition which develops when the reflux of stomach contents cause troublesome symptoms and/or complications.At present,more than half the patients with GERD symptoms were diagnosed as having nonerosive reflux disease(NERD).However,by careful analysis,the majority of NERD patients did not have completely normal endoscopic finding but were found to have subtle distal esophageal mucosal changes.Forty-eight patients with suspected minimal change esophageal reflux disease(positive GerdQ but normal conventional endoscopy)and forty asymptomatic control were recruited.The new LCI(GF-L590WR) was performed.The criteria for positive liquid crystal thermography (LCT) were:a)triangular indentation,b)punctuate erythema.

ELIGIBILITY:
Inclusion Criteria:

* age more than 18 year old
* ability to provide written informed consent and undergoing an upper endoscopy
* no PPI therapy in previous 2 weeks and no esophageal tumor or stenosis or history of esophageal surgery
* Patients with more than 3 reflux episodes/week and absence of mucosal breaks at conventional endoscopy，The PPI test was positive

Exclusion Criteria:

* unable to provide informed consent
* erosive esophagitis or diagnosis of erosive esophagitis within the recent 6 months
* presence of columnar lined epithelium
* evidence of cancer or mass lesion in the esophagus, gastric lesions (ulcer, polyp, cancer)
* previous gastrointestinal surgery
* esophageal strictures
* chronic use of medications known to affect esophageal motility
* presence of systemic diseases that might interfere with esophageal motility
* use of proton pump inhibitors(PPI) or histamine2-receptor antagonists in the last 4 weeks

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients undergoing an outpatient endoscopy
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2017-01-15 (Actual); Primary Completion 2017-10-30 (Estimated); Study Completion 2017-12-30 (Estimated)

PRIMARY OUTCOMES:
observation minimal change esophagitis | 5 months
  conducted to assess the effectiveness of LCI for diagnosing esophageal MCE when compared to conventional white-light endoscopy (WLI).Meanwhile， interobserver and intraobserver variation in the use of LCI system between endoscopists with different levels of experience.

SECONDARY OUTCOMES:
Improvement observation agreement of Los Angeles classification system for GERD using LCI by comparing with that under white endoscopy | 5 months
  It is anticipated that the use of Linked Color Imaging(LCI) will significantly improve the observation agreement of Los Angeles Classification when detected as opposed to White-light endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Yan Liu, Ph.D., Principal Investigator — Affiliate Hospital to Academy of Military Medical Sciences
Locations (1):
- Department of gastroenterology,Affiliated Hospital to Academy of Military Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sharma P, Wani S, Bansal A, Hall S, Puli S, Mathur S, Rastogi A. A feasibility trial of narrow band imaging endoscopy in patients with gastroesophageal reflux disease. Gastroenterology. 2007 Aug;133(2):454-64; quiz 674. doi: 10.1053/j.gastro.2007.06.006. Epub 2007 Jun 8. PMID 17681166
- [Result] Wang WH, Tsai KY. Narrow-band imaging of laryngeal images and endoscopically proven reflux esophagitis. Otolaryngol Head Neck Surg. 2015 May;152(5):874-80. doi: 10.1177/0194599814568285. Epub 2015 Jan 27. PMID 25628366
- [Result] Lei WY, Liu TT, Yi CH, Chen CL. Disease characteristics in non-erosive reflux disease with and without endoscopically minimal change esophagitis: are they different? Digestion. 2012;85(1):27-32. doi: 10.1159/000334715. Epub 2011 Dec 13. PMID 22156539
- [Derived] Deng P, Min M, Dong T, Bi Y, Tang A, Liu Y. Linked color imaging improves detection of minimal change esophagitis in non-erosive reflux esophagitis patients. Endosc Int Open. 2018 Oct;6(10):E1177-E1183. doi: 10.1055/a-0602-3997. Epub 2018 Oct 8. PMID 30302374